CLINICAL TRIAL: NCT06714760
Title: Evaluation of the Galea-pericranium Flap in Reconstruction of Oral Cavity Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMF-PC22
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Oral Disease
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient (Experimental): The study will involve patients referred to the Department of Maxillofacial Surgery, IRCCS Azienda Ospedaliero-Universitaria di Bologna who require simple reconstruction following parcellar resections of the mandibular gingival region. It is planned to recruit during the above period 5 patients who meet the following inclusion and exclusion criteria.
  Interventions: Procedure: Reconstruction following parcellar resections of the mandibular gingival region

INTERVENTIONS:
Procedure: Reconstruction following parcellar resections of the mandibular gingival region — In our surgical approach, we have used periosteum, galea, or pericranium flaps for reconstruction of bone and tissue defects in the cervicofacial region, with excellent results. To treat mandibular osteoradionecrosis, we harvested periosteum flaps from the radius, demonstrating efficacy in bone regeneration. For minor defects, such as those of the nose, we used flaps from the medial femoral condyle, despite the complexity of harvesting.
  The cranial region, particularly the temporo-parietal area, offered excellent vascularization, allowing the use of revascularized flaps for reconstruction of the oral mucosa after removal of carcinomas. These flaps have also been effective in the treatment of pharyngeal fistulas, proving to be a functionally reliable solution for oral cavity and cervicofacial defects.

SUMMARY:
The overall objective of this study is to evaluate the safety of using the galea and pericranium (fascio-periosteal) temporal flap in the reconstruction of mandibular gingival defects.

DETAILED DESCRIPTION:
Reconstruction with free flaps is a routine practice in head and neck surgery because of better functional, aesthetic results and generally higher success rates.

Current applications of this practice include reconstructive surgeries that follow excisions of neoplastic lesions involving the oral cavity. Following resection of the primary tumor, reconstructive surgery is usually necessary in order to restore function to the oral cavity.

The most appropriate reconstructive method is determined by several factors, including the characteristics of the defects and primary tumor site, the general medical condition, the patient's social history, the prognosis, and the surgeon's expertise. Reconstructive methods usually follow a "reconstructive ladder," starting with a skin graft and ending with a microvascular free flap.

Free tissue transfers are currently one of the most popular and reliable techniques for oral reconstruction.

The use of periosteal flaps for reconstruction of bone defects has been described by several authors. In particular, a well-known technique by Bettoni et al. [5] demonstrated excellent results, also in terms of bone regeneration, following the use of free periosteum flaps taken from radius in the treatment of osteoradionecrosis of mandible.

Free flaps of periosteum and osteoperiosteum of the medial femoral condyle have also been widely used for minimal bone reconstructions, such as those of the nasal bone, again with excellent results . However, harvesting these flaps is complex and the periosteum obtained is small in size.

Based on the assumption that the cranial region would provide surgeons with more options in terms of harvesting periosteum flaps to reconstruct soft and hard tissue defects, previous clinical experiences have explored the possibility of harvesting a galea and pericranium flap for reconstruction of oral mucosal defects resulting from excision of squamous cell carcinomas, obtaining positive results. Indeed, the temporal region is an important donor site in reconstructive surgery of the head and neck region, from which pedicled flaps of muscle, fascia, and skin can be harvested.

In particular, the vascular supply of the pericranial temporo-parietal region was evaluated in the above experience.

Previous clinical experience has demonstrated the efficacy of such a flap, used for the treatment of pharyngeal fistulas, as a revascularized free graft.

In conclusion, this type of flap has been shown to be functionally reliable for defects of the cervicofacial district, so we propose to apply it to parcellar defects of the oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years;
* Patients with mandibular gingival defects involving the anterior or lateral aspect of the mandible;
* Patients in whom basal structural integrity of the mandibular bone is maintained;
* Patients with a minimum follow-up of 3 months;
* Obtaining informed consent.

Exclusion Criteria:

• Patients with history of previous surgery that bilaterally altered the superficial temporal vasculature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-01-11 (Estimated); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
outcomes | 18 months
  Number and % of patients with adequate flap viability, defined as effective vascular supply and complete rooting of the flap at the recipient site, without tissue necrosis. Partial viability will be considered as incomplete rooting of the flap with associated peripheral tissue necrosis affecting less than 1/3 of the surface de

CONTACTS AND LOCATIONS:
Overall Officials: Achille Tarsitano, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS - Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna, Italy